CLINICAL TRIAL: NCT03378700
Title: Evaluation on the Effects of a Brief Hope Intervention to the Decision Making in the Chinese Chronic Kidney Disease Patients on Their Management Options: a Randomised Controlled Trial
Brief Title: Effects of a Brief Hope Intervention to the Decision Making
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS2018
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD; Hope Intervention; decision making
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a single-blinded randomised controlled trial. On completion of the baseline assessment and the screening procedure, eligible participants will be randomly assigned in equal number into either a brief hope intervention (BHI) or the control group using sets of computer-generated random numbers.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator and the nurse providing the intervention are aware of the patient group assignment. Assessment of the baseline and endpoints of the patient outcomes will be performed by an independent research assistant blinded to group allocation, who was not involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Hope Intervention Group (Experimental): In addition to the pre-dialysis educational programme on self-care and treatment options for ESRF patients as per the control group, brief hope intervention will be offered: a four-weeks individual intervention. Two face-to-face sessions (1-hour) and two telephone follow up sessions (30 minutes) in between. A booklet modified from the goal worksheet in Lopez et al. (2000) will be prepared for the participants for reviewing their planned goals, recording achieved targets and successful experiences.
  Interventions: Behavioral: Brief Hope Intervention
- Pre-dialysis Education Group (Active Comparator): Pre-dialysis educational class and standard care such as clinic follow up and normal hospital care will be provided. This session is led by clinicians with renal nursing training. The educational class aims at providing information on the treatment modalities for patients with ESRD, signs and symptoms of their illness and the basic advice on the importance of adherence to healthy lifestyle, nutrition and medications. Logistic call and social communication will be offered and initiated by trained nurses in the second week and the third week
  Interventions: Other: Pre-dialysis Education Group

INTERVENTIONS:
Behavioral: Brief Hope Intervention — The present Brief Hope Intervention (BHI) is a four-weeks individual intervention, consisting of four sessions: two face-to-face sessions (1-hour) and two telephone follow up sessions (30 minutes) in between.
  The facilitator will guide participants to imagine how they navigate themselves to circumvent possible obstacles and accomplished their set goals and experience positive emotions.
  A booklet will be given to the participants for reviewing their planned goals, recording achieved targets and successful experiences.
  Arms: Brief Hope Intervention Group
Other: Pre-dialysis Education Group — Pre-dialysis educational class and standard care such as clinic follow up and normal hospital care will be provided. This session is led by clinicians with renal nursing training. The educational class aims at providing information on the treatment modalities for patients with ESRD, signs and symptoms of their illness and the basic advice on the importance of adherence to healthy lifestyle, nutrition and medications. Logistic call and social communication will be offered and initiated by trained nurses in the second week and the third week
  Arms: Pre-dialysis Education Group

SUMMARY:
Introduction A Hong Kong study found that more than half of the chronic kidney disease (CKD) patients declined peritoneal dialysis (PD) and preferred receiving palliative care, although PD is vital for early preservation of residual kidney functions. Decision-making was found to be influenced by feelings of hopelessness, leading to underestimation and the pursuit of a successful plan of action. Cumulative evidences revealed that hope is a factor that heightens positive expectations in patients, and could lead to consideration of wider alternatives and thorough decision making.

Aim The aim of this study is to examine the effectiveness of a brief hope intervention in reducing the decisional conflict and improving the quality of life of CKD patients who have to plan for receiving dialysis therapy. If patients' quality of decision-making could be improved, timely initiation dialysis and less decisional regret is expected.

Method This study is a single-blinded randomised controlled trial. On completion of the baseline assessment and the screening procedure, eligible participants will be randomly assigned in equal number into either the experimental group (education programme plus a brief hope intervention) or the control group (education programme) using sets of computer-generated random numbers.

Patients attending the outpatient renal clinic of a regional hospital in HK will be approached. Stage 5 CKD patients (GRF equal to or less than 15) who are planned to receive dialysis therapy or palliative care will be invited to join the study. Taking into consideration of attrition and the health status of the palliative care patients, it was appropriate to sign up 36 participants per arm, correlation alpha value 0.6, 0.5 effect size with a power of 0.70.

There are four waves of data collection, which will be done before the commencement of the intervention (T1), immediately post-intervention (T2) and one month (T3) and three months (T4) after the completion of programme. Primary Outcomes include the assessing the patients' decisional conflict, strength of preference, on their choice of treatment modalities between peritoneal dialysis and palliative care, and health resources utilization. Secondary outcomes measure hope level change and quality of life. Sociodemographic and socioeconomic information will be collected. Two open-ended questions will be used to explore the perceived impact and benefits of the intervention.

DETAILED DESCRIPTION:
Decision Making in Patients with Chronic Kidney Disease Patients with chronic kidney disease (CKD) stage 5 (estimated creatinine clearance equal to or less than 15 mL/min/1.73 m2), would face tough decisions on their treatment options when they were discovered to have end stage renal disease (ESRD), as their decisions affected their long term QoL. In general, when patients reach stage 4 CKD, taking into the account of the other symptoms and complications, dialysis initiation would be discussed. Peritoneal dialysis (PD) first policy has been adopted in the Hong Kong public health care system since 1985. It showed comparable patient survival outcomes to haemodialyis and early preservation of residual kidney functions. Nonetheless, a Hong Kong study found that more than half of these patients declined PD and preferred receiving palliative care. For those who decided to have conservative treatment may require urgent dialysis when their symptoms deteriorated such as dyspnoea. These patients may have decisional regret and would like to revert their initial choice. As such, helping patients to rigorously consider their preferences and concern is crucial.

Quality Decision Making Decision-making to commence or decline renal therapy in ESRD is a complex and dynamic process and evolves over time. It was found that planned dialysis in predialytic stage of CKD could reduce hospitalization duration, economic costs, mortality and improves QoL and depression. Standard pre-dialysis consultations, providing information on comparative risks, benefits and alternatives appeared inadequate to guide individualized decisions that are affected by personal values and perceptions. In a similar vein, a randomised control trial on asymptomatic abdominal aortic aneurysm on increasing patients' knowledge about the disorder and better informed them about elective surgery or watchful waiting did not reduce decisional conflict. Despite good knowledge, irrational choices were made. Patients felt that they have autonomy and were offered a treatment alternative if the consultation stimulated them to think of additional questions before making a decision. Some patients tried to take control of their progressive status of renal failure, while others tried to take control of their emotions. Determining the patients' readiness and facilitating patients to express their struggles to make value congruent decisions require more than a health education. Subsequent motivation after nephrology consultation become a vital step to enable these patients to initiate planned dialysis.

The Importance of Hope to Quality Decision Making Hope theory is adopted as the framework in the present study, where hope was believed as the central agent to facilitate the change process. By increasing hope level, the likelihood of therapeutic change will be increased. It is hypothesized that increasing hope would lead to selecting PD as recommended, stronger decision to the treatment, less decisional conflict and reduced emergency room visits or hospitalisation . Patients facing chronic illnesses would lead to psychological stress, anxiety, depression, fear and hopelessness. Prognostic uncertainty, subjective perception of a worsening health status, experience of quality of life, and even a sense of abandonment were expressed in the patients with chronic kidney diseases. Both depression and hopelessness was documented in renal failure patients. In a systematic review, cognitive appraisal was also found to have the largest effect size that associate with depression in patients with ESRD. Another systematic review and thematic synthesis also revealed five themes of concerns; (1) invasive suffering, such as loss of independence, treatment burden and harm, (2) personal vulnerability such as autonomy and dignity, (3) relational responsibility, for instance, protecting others from grief, (4) existential tensions such as preserving self-identity, and (5) preparedness, for example, decisional clarity, spirituality and hope. As such, both cognitive and emotional strategies should be integrated to facilitate effective decision making.

Despite the mechanisms by which positive emotions impact on decision making are not clearly understood, it was found that positive affect leads to efficient and thorough decision-making , that applied to physician's diagnostic process. It has been found that hope is one of the diverse positive emotions, which could lead to consideration of wider alternatives. Thus, it may lead to a more thorough exploration of the treatment options and consequences during the decision making process. Evidence has shown that high-hope individuals were found to be more creative and effective problem solvers. It is timely to translating these findings to wider clinical perspectives to enhance quality decision-making. Whether improving the hopeful state of patients with ESRF would lead to decrease decisional conflict or regrets remains under explored. Investigating whether improving the hopeful state of CKD patients would lead to better health outcomes will advance the application of hope in clinical interventions. The present study aimed to investigate the effect of brief hope therapy on the patients with stage 5 CKD when renal dialysis is recommended.

Hope Intervention Hope therapy that based on Snyder's conceptualization of hope is adopted in the present study. Three core features: (1) goal setting (goals), (2) problem solving (pathways) and (3) positive self-talk (agency), underlie the key hope strategies used in the intervention. Hope therapy is delivered within the principles of cognitive behavioural therapy (CBT), but its focus complemented the traditional CBT by shifting the primary focus on positive potentials, thereby promoting meaning in life, fostering personal strengths and positive changes. Despite the controversy about hope interventions lies on being overly optimistic is harmful, nurturing hope was found to be one of the significant elements in staying positive in the coping experiences of Chinese cancer patients. More importantly, hope is a pursuit toward a desirable future openness to possibilities, affirmation and reflection about one's capacity to reach self-established goals, and engagement in actions to make a difference in the outcome.

ELIGIBILITY:
Inclusion Criteria:

The candidates should meet the below criteria will be recruited.

1. age ≥ 18 years
2. clinically diagnosed to have End Stage Renal Diseae (ESRD) and Glomerular Filtration Rate (GFR) less than or equal to 15
3. willing to participate in face-to-face activities and telephone follow up
4. alert and oriented, able to sustain for approximately one hour of attention and interaction
5. communicable in Cantonese, able to read and write Chinese
6. could be reached by phone

Exclusion Criteria:

Patients having one or above of the below conditions will be excluded from the study.

1. patients who have been receiving renal replacement therapy
2. patients who have failed kidney transplant
3. patients who are unable to communicate in Cantonese
4. patient who has hearing deficit
5. Patient who are disoriented, delirious or cognitively impaired
6. patients who are clinically depressed diagnosed by medical doctors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Decision Making Profile and Decisional Conflict Scale (DCS) | 3 months
  The scale was recommended in Shared Decision-making Programme of the U.K. National Health Services (National Health Service & Capita Group, 2012). It is a 16-items tool that consists of five subscales rated on a 5-point Likert scale. Reliability of DCS is good (Cronbach's alpha = .78) and construct validity discriminating between known groups (effect size .4-.8), and responsiveness to change is good in studies of decision supporting interventions (ES .4-1.2) (O'Connor, 2010).

SECONDARY OUTCOMES:
Strength of Preference (SP) | 3 months
  This is a single item, 4 point Likert scale, ranging from 1 (weak preference) to 4 (very strong preference), that measures the strength of preferred treatment option (Stalmeier & Roosmalen, 2009). A value of zero was designated to indicate 'undecided'.
State Hope Scale (SHS) | 3 months
  The SHS Chinese version (Mak, Ng, & Wong, 2011) is a self-report instrument consisting of 6 items (Snyder et al., 1996) used to assess the two ongoing hope indices related to the pathways and agency of hopeful thinking. It is rated on an 8-point scale with 1 = definitely false and 8 = definitely true. Cronbach's alpha for these two subscale items ranged from 0.74 to 0.93 (all ps < 0.001).
Kidney Disease Quality of Life Questionnaire (KDQOL-36) Cantonese Chinese Version | 3 months
  This self-reported disease-targeted instrument is specific for assessing the health-related QoL of CKD patients (Chow & Tam, 2014). It comprises of three subscales (24 items): (1) Symptoms and Problems (12 items), (2) Burden of Kidney Disease (4 items), and (3) Effects of Kidney Disease (8 items). Another 12 items were adopted from the Short Form Health Survey (SF12), which comprises of two sub-scores of Physical Component Summary (PCS) and Mental Component Summary (MCS). The higher the scores indicating better QoL. The Chinese version reported an overall internal consistency ranged from 0.72-0.94, while the intra-class correlation (ICC) test-retest reliability is 0.81-0.96 in the various domains (Tao, Chow, & Wong, 2014).
Healthcare Resource Utilisation Data | 3 months
  This profile reflects the complex and dynamic situation of QoL in CKD participants.
  Three health services utilization indicators will be collected for a period of three months to determine their association with the subjective measures.
  1. the number of hospital readmissions (number of times within 30 days after discharge),
  2. emergency room visits (the lower the number, the lesser the need),
  3. recommended treatment choice, patients' initial and final treatment choice
  4. refusal to dialysis initially and reverting to dialysis from palliative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kitty Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan K, Wong FKY, Tam SL, Kwok CP, Fung YP, Wong PN. Effectiveness of a brief hope intervention for chronic kidney disease patients on the decisional conflict and quality of life: a pilot randomized controlled trial. BMC Nephrol. 2022 Jun 14;23(1):209. doi: 10.1186/s12882-022-02830-7. PMID 35701732